CLINICAL TRIAL: NCT06197152
Title: Identification and Clinical Validation of Biomarkers Associated With Clinical Severity in Adults Infected With Respiratory Syncytial Virus
Brief Title: Identification and Clinical Validation of Biomarkers Associated With Clinical Severity in Adults Infected With RSV
Acronym: ARF-RSV
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221290
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus; RSV; Respiratory infection; Febrile acute respiratory syndrome; Immuno-virological determinants
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal samples will be obtained sequentially (i.e., at day 0, day 3-4, day 5-7, and day 14 of inclusion) for virological and transcriptomic analyses. Blood samples will also be collected at day 0 (EDTA tubes and Paxgene tubes), day 5-7, and day 14 for peripheral transcriptomic analyses and plasma banking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 100 patients with RSV diagnosis: Patients with acute respiratory infection and positive nasopharyngeal PCR or other respiratory specimen for RSV.
  Interventions: Other: Nasopharyngeal swabs and biological collection
- 33 control patients: Patient admitted for acute respiratory syndrome with no diagnosis of respiratory infection or immunosuppression.
  Interventions: Other: Nasopharyngeal swabs and biological collection

INTERVENTIONS:
Other: Nasopharyngeal swabs and biological collection — * Nasopharyngeal PCR
  * Blood and virological samples taken as part of the research will be included in a biological collection

SUMMARY:
A short description, 5000 characters Intro: Respiratory Syncytial Virus (RSV) is a frequent, ubiquitous agent of respiratory viral infections. It is the leading viral cause of lower respiratory tract infection (LRTI) in infants and also causes significant morbidity and mortality in adults, especially in the elderly, in patients with cardiorespiratory comorbidities [e.g., patients with Chronic Obstructive Pulmonary Disease (COPD) and/or heart failure], and in immunocompromised patients. Clinical phenotyping of RSV respiratory infections has shown that the occurrence of LRTI in RSV-infected patients is associated with the need for ventilatory support and an increased risk of mortality. Virological data also suggest that there is a relationship between high nasopharyngeal viral replication levels and a poor prognosis, although these data have not been confirmed in other studies. Beyond viral load, the impact of viral subtypes on the severity of RSV infection is controversial. Few data have explored the prognostic value of genetic diversity (i.e., role of RSV variants, mutations occurring during clinical course) in RSV-infected adult patients with acute respiratory failure.

Objective: The main goal of the present study is to identify and validate biomarkers associated with RSV severity in adults infected with RSV that will be useful to guide treatment decisions in the future. This study will additionally characterize the thus far unknown genetic diversity of RSV in hospitalized adults with severe and mild infections, in order to anticipate virological escape mechanisms from current and future treatments.

Method: This is a prospective multicenter cohort study of patients with RSV infection admitted to the hospital. These patients will be followed-up for 28 days. Nasopharyngeal samples will be obtained sequentially (i.e., at day 0, day 3-4, day 5-7, and day 14 of inclusion) for virological and transcriptomic analyses. Blood samples will also be collected at day 0 (EDTA tubes and Paxgene tubes) for peripheral transcriptomic analyses and plasma banking.

The 100 first patients included in the study will be allocated to the development cohort and the last 100 patients will be allocated to the validation cohort.

ELIGIBILITY:
Group of patients with RSV diagnosis

Inclusion Criteria:

* Age > 18 years
* Positive RSV RT-PCR in nasopharyngeal swab
* Patient admitted to the hospital (intensive care unit or medical ward admission at inclusion) with clinical signs of lower respiratory tract infection (defined as the presence of two or more respiratory signes (cough, dyspnea, sputum production, wheezing, tachypnea (respiratory rate>20/min) or one respiratory sign plus one or more systemic symptoms (fatigue and fever)) requiring hospitalization.
* No objection letter (from the patient or a member of family if the patient is not physically able to give consent

Exclusion Criteria:

* Co-infection with other respiratory viruses
* Persons under guardianship/guardianship
* AME (state medical aid) patient

Group of "control" patients

Inclusion Criteria :

* Age>18 years
* Patient's consent
* Enrolled in a social security plan
* Admitted for an acute respiratory syndrome
* No diagnosis of respiratory infection in the 4 weeks prior to inclusion
* Negative RSV nasopharyngeal PCR (or other respiratory specimen) collected within the last 48 hours
* No immunosuppression (HIV infection, bone marrow or solid organ transplantation, post-chemotherapy aplasia, immunosuppressive therapy, corticosteroid therapy (> 200 mg/d hydrocortisone or equivalent within 4 weeks prior to inclusion)

Exclusion Criteria :

* Persons under guardianship/guardianship
* AME (state medical aid) patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RSV diagnosis : Patients hospitalized for RSV respiratory infection requiring hospital admission.
  Control group : patients admitted for acute respiratory failure free for RSV or any other infection.
Sampling Method: Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory and immune response | within 72h of hospitalization
  Patients with severe disease, defined as developing acute respiratory failure with a World Health Organization (WHO) ten-point scale ≥6 at any time of hospital stay, and those with mild disease (WHO ten-point scale remaining <6 during hospital stay) will be compared using several biological tools, in particular the inflammatory and immune response assessed by transcriptomic analyses in peripheral blood and in respiratory samples (nasopharyngeal swabs and bronchoalveolar lavage fluid or tracheal aspirates when available).

SECONDARY OUTCOMES:
Inflammatory and immune response during hospital stay | during hospitalization (until day 28).
  Differences between the two groups of RSV-infected patients, with severe disease (WHO ten-point scale ≥6) versus mild disease (WHO ten-point scale remaining <6), of inflammatory and immune responses assessed by transcriptomic analyses in respiratory samples (nasopharyngeal swabs and bronchoalveolar lavage fluid or tracheal aspirates when available).
RSV genetic variability during hospitalization | during hospitalization (until day 28)
  Relationship between viral level dynamics and intra-individual viral genetic variability in respiratory samples (nasopharyngeal swabs and bronchoalveolar lavage fluid or tracheal aspirates when available).
RSV genetic variability at admission | during hospitalization (within 72h of hospitalization)
  Differences between the two groups of RSV-infected patients, with severe disease (WHO ten-point scale ≥6) versus mild disease (WHO ten-point scale remaining <6), of inter-individual viral genetic variability in respiratory samples (nasopharyngeal swabs).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-André Natella, PhD, Study Chair — APHP URC
Locations (1):
- Intensive Care Unit Henri Mondor APHP, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION